CLINICAL TRIAL: NCT07385482
Title: Impact of Chronic and Acute Cardiovascular Diseases in Older Intensive Care Patients: A Prospective Multicenter Observational Study - VIP4
Brief Title: Chronic and Acute Cardiovascular Diseases in Elderly Intensive Care Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: VIP4
Record Dates: First submitted 2026-01-20; First posted 2026-02-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Chronic Cardiovascular Disease; Acute Cardiovascular Disease; Frailty
Keywords: older intensive care patients; intensive care unit; cardiovascular disease; frailty; multimorbidity; mortality; functional outcome; health-related quality of life
MeSH Terms: conditions — Frailty; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Very old patients are a rapidly growing and vulnerable population in acute cardiovascular care but remain underrepresented in clinical trials. Clinical outcomes in older intensive care unit (ICU) patients are determined less by chronological age than by their clinical phenotype, including cardiovascular comorbidities, frailty, polypharmacy, and functional and cognitive impairment. This prospective multicenter observational study aims to assess the impact of chronic and acute cardiovascular diseases on long-term outcomes and functional trajectories in older ICU patients. Using the international VIP research network, approximately 4,000 patients will be enrolled across different ICU specialties and healthcare systems and assessed multidimensionally using validated clinical scores. The study seeks to improve risk stratification and outcome prediction in older critically ill patients with cardiovascular disease and to address existing evidence gaps in acute cardiovascular and intensive care medicine.

DETAILED DESCRIPTION:
The primary aim of this prospective multicenter observational study is to investigate the impact of chronic and acute cardiovascular diseases on the clinical phenotype, short-term outcomes, and long-term functional trajectories of older intensive care unit (ICU) patients. The main hypothesis is that patients with chronic or acute cardiovascular diseases differ in their pre-ICU clinical phenotype and have a higher risk of adverse short-term outcomes and impaired long-term functional recovery compared with patients without these conditions. Using the established international VIP research network, older ICU patients will be assessed multidimensionally using validated instruments and routinely collected clinical data across different ICU specialties (cardiac, cardio-surgical, internal medicine, and surgical ICUs) and healthcare systems.

The primary endpoint of the study is 6-month all-cause mortality. Secondary endpoints include functional status and health-related quality of life during follow-up.

Pre-existing comorbidities will be captured using the AHRQ Elixhauser Comorbidity Index, with detailed documentation of chronic cardiovascular comorbidities and medication history. Frailty and functional status will be assessed using the Clinical Frailty Scale and the Katz Index, while baseline cognitive function will be evaluated using the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE). Health-related quality of life prior to the acute illness will be assessed using the EQ-5D-5L. Nutritional status will be evaluated using the Geriatric Nutritional Risk Index (GNRI) and the Global Leadership Initiative on Malnutrition (GLIM) criteria (e.g. body weight and dietary history) At ICU admission and during the ICU stay, routinely available laboratory parameters including albumin, lactate, international normalized ratio (INR), HbA1c, and hemoglobin will be recorded. Disease severity will be assessed using the Sequential Organ Failure Assessment (SOFA) score at admission and during follow-up. Data on ICU interventions, including invasive mechanical ventilation, vasopressor therapy, renal replacement therapy, mechanical circulatory support, enteral and parenteral nutrition, and physiotherapy, will be documented. Hemoglobin levels at ICU admission and discharge as well as the highest and lowest values during the ICU stay will be captured.

Approximately 4,000 patients are planned to be enrolled within 12 months, allowing predefined subgroup analyses according to age, sex, frailty status, and cognitive function using advanced exploratory analytical approaches. The study aims to contribute to closing the existing evidence gap regarding chronic and acute cardiovascular disease in older critically ill patients

ELIGIBILITY:
Inclusion Criteria:

* 80 years or older
* Admission to the intensive care unit
* Signed informed consent or absence of discernible indications suggesting the presumed intention of the patient not to participate in the study.

Exclusion Criteria:

* < 80 years
* Absence of informed consent
* Discernible indications suggesting the presumed intention of the patient not to participate in the study.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study focuses on older intensive care unit patients with chronic and acute cardiovascular diseases and is coordinated across multiple international sites using standardized data collection procedures.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
mortality | within 6 months
  surivival or death

SECONDARY OUTCOMES:
Functionality and Quality of Life | 6 months
  measured by clinical fraility scale: Scores range from 1 (Very Fit) to 9 (Terminally Ill). Higher scores indicate greater frailty and worse health status
Functionality and Quality of Life | 6 months
  measured by katz acitivies of daily living (assessment of ability to perform daily activities): Scores range from 0 to 6, with higher scores indicating greater independence and better functional status
Functionality and Quality of Life | 6 months
  measured by EQ-5D-5L (assessment of health-related quality of life): Individual response patterns will be reported as EQ-5D-5L health states (e.g., 11111 indicating no problems in all five dimensions), allowing a descriptive assessment of dimension-specific limitations
Long-term survival and readmission rate | up to 12 months
  Long-term survival and readmission rate

OTHER OUTCOMES:
The combined endpoint aims to evaluate both survival outcomes and functional independence | 6 months
  Survival, Improvement or stability in frailty status according to the Clinical Frailty Scale compared to baseline, Improvement or stability in the ability to perform daily activities according to the Katz Activities of Daily Living compared to baseline, Improvement or stability in health-related quality of life according to the EQ-5D-5L compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, MD, Study Chair — Division of Cardiology, Pulmonary Disease and Vascular Medicine at University Hospital Duesseldorf; Christian Jung, MD, Principal Investigator — Division of Cardiology, Pulmonary Disease and Vascular Medicine at University Hospital Duesseldorf
Locations (1):
- University Hospital Duesseldorf, Düsseldorf, Germany